CLINICAL TRIAL: NCT01248507
Title: Comparative Evaluation of COPD Specific Quality of Life Assessment Questionnaires (the COPD Assessment Test, the Clinical COPD Questionnaire, the COPD Severity Score and the Airways Questionnaire 20 as Predictive Tools for Risk of Acute COPD Exacerbations
Brief Title: Predictive Questionnaires for Risk of Acute COPD (Chronic Obstructive Pulmonary Disease) Exacerbations
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: RO-2455-401-ES; NYC-EPOC-2009-01; U1111-1146-5711 (Registry Identifier: UTN (Who))
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
COPD patients frequently suffer intermittent exacerbations of their disease characterised by acute deterioration of symptoms. Acute exacerbations of COPD (AECOPD) are associated with significant impairment of health status, use of health care resources, poor prognosis and increased mortality. The development of simple and practical predictive tools would help to identify COPD patients at greater risk of suffering exacerbations, which is important since those patients would need more intense and early treatment.

This one-year prospective cohort non-drug study will evaluate several COPD-specific questionnaires as predictive tools and the presence of cardiovascular comorbidities as risk factors, for the composite events in study cohorts. The trial duration consists of a screening period (4-6 weeks) and a follow-up period (12 months), 4 visits in total along the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 40 years
* Patients fulfilling criteria for COPD according to the Global initiative for chronic obstructive pulmonary disease (GOLD) stage I or higher
* Smokers or ex-smokers of at least 10 pack-years
* Patients suffering an AECOPD either:

  1. Admitted to hospital due to AECOPD (severe exacerbation) or
  2. Confirmed AECOPD at GP (general practitioner) setting (moderate exacerbation) Definition AECOPD: Increase in respiratory symptoms requiring treatment with oral corticosteroids, antibiotics or both.

Exclusion Criteria:

* Patients who have never smoked
* Patients with active long-term respiratory disease (e.g. bronchial asthma, cystic fibrosis, severe bronchiectasis, malignancy, restrictive lung diseases etc.)
* Exacerbation of COPD due to other causes such as pneumothorax and acute decompensated congestive heart failure
* Difficulties in communication (cognitive deterioration, sensorial disability, language barriers)
* Severe disease with poor vital prognosis (life length expectancy less than one year)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 634 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Comparative evaluation of the predictive value of the COPD Assessment Test (CAT), Clinical COPD Questionnaire (CCQ), COPD Severity Score (COPDSS) and the Airways Questionnaire 20 (AQ20) questionnaires (in hospital) | one year
  Comparative evaluation of the predictive value of the CAT, CCQ, COPDSS and the AQ20 questionnaires for the composite event of mortality and re-hospitalization for COPD, in a one year follow-up of a cohort of COPD patients admitted for an exacerbation, enrolled in hospital.
Comparative evaluation of the predictive value of the CAT, CCQ, COPDSS and the AQ20 questionnaires (in primary care) | one year
  Comparative evaluation of the predictive value of the CAT, CCQ, COPDSS and the AQ20 questionnaires for the composite event of any exacerbation, mortality and hospitalization for COPD, in a one-year follow-up of a cohort of COPD patients enrolled in primary care.

SECONDARY OUTCOMES:
To evaluate cardiovascular comorbidities as risk factors for the composite events in the hospital and the primary care cohorts. | one year

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Nycomed Pharma S.A., Madrid, Spain